CLINICAL TRIAL: NCT02733042
Title: A Phase 1/2, Open-label, Multi-center Study to Assess the Safety and Tolerability of Durvalumab (Anti-PDL1 Antibody) as Monotherapy and in Combination Therapy in Subjects With Lymphoma or Chronic Lymphocitic Leukemia
Brief Title: A Study to Determine Dose, Safety, and Efficacy of Durvalumab as Monotherapy and in Combination Therapy in Subjects With Lymphoma or Chronic Lymphocytic Leukemia
Acronym: FUSION NHL 001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-NHL-001; 2015-003516-21 (EudraCT Number)
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Lymphoma; Chronic Lymphocytic Leukemia; Durvalumab; Anti-PD-L1 Antibody; MEDI4736; Immune Checkpoint; Lymphatic Disease; B-Cell Malignancies; Abscopal Effect; Lenalidomide; Bendamustine; Rituximab; Ibrutinib; Lymphoma, B-Cell; Lymphoma, Non Hodgkin,; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell,; Lymphoma, Follicular; Lymphoma, Diffuse Large B-Cell; Lymphoma, Mantle Cell; Lymphoma, Small Lymphocytic; Immune System Diseases; Immunoproliferative Disorders; Lymphoproliferative Disorders
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphatic Diseases; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Immune System Diseases; Immunoproliferative Disorders; Lymphoproliferative Disorders | interventions — durvalumab; Lenalidomide; Rituximab; ibrutinib; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Within Arms A, B, and C participants on the dose-finding part were enrolled sequentially according to a 3+3 design. All treatment arms were to be open for enrollment at study start except in the US, where Arm D was to enroll depending on the availability of treatment slots and following the completion of assessment of responses from the combination therapy arms.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A: Durvalumab + Lenalidomide ± Rituximab (Experimental): Participants assigned to Arm A will receive:
  * Durvalumab 1500 mg intravenous (IV) infusion on Day 1 of Cycles 1 through 13 (ie, 12 months) and
  * Lenalidomide orally at assigned dose levels (10 mg, 15 mg or 20 mg) once daily on Days 1 to 21 of:
    * Cycles 1 through 13 in indolent non-Hodgkin's lymphoma (NHL) or
    * All cycles of treatment period until disease progression, unacceptable toxicity, or discontinuation for any other reason in aggressive NHL
  * Rituximab 375 mg/m² IV infusion every week in Cycle 1 (Days 2, 8, 15, 22) and on Day 1 of Cycles 2 through 5.
  All treatment cycles were 28 days.
  Interventions: Drug: Durvalumab; Drug: Lenalidomide; Drug: Rituximab
- Arm B: Durvalumab + Ibrutinib (Experimental): Participants assigned to Arm B will receive:
  * Durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13
  * Ibrutinib orally at assigned dose levels (280 mg, 420 mg, or 560 mg) once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
  All treatment cycles were 28 days.
  Interventions: Drug: Durvalumab; Drug: Ibrutinib
- Arm C: Durvalumab + Rituximab ± Bendamustine (Experimental): Participants assigned to Arm C will receive:
  * Durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13
  * Rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6 (for CLL the rituximab dose will be 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose)
  * Bendamustine IV infusion at assigned dose levels (70 mg/m² or 90 mg/m²) on Days 1 and 2 of Cycles 1 through 6.
  All treatment cycles were 28 days.
  Interventions: Drug: Durvalumab; Drug: Rituximab; Drug: Bendamustine
- Arm D: Durvalumab Monotherapy (Experimental): Participants assigned to Arm D will receive durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13. All treatment cycles were 28 days.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Administered as an IV infusion (250 mL) over approximately 1 hour in duration
  Other Names: MEDI4736; IMFINZI®
Drug: Lenalidomide — Administered orally
  Other Names: Revlimid®
  Arms: Arm A: Durvalumab + Lenalidomide ± Rituximab
Drug: Rituximab — Administered by intravenous infusion
  Other Names: Rituxan®; MabThera®
  Arms: Arm A: Durvalumab + Lenalidomide ± Rituximab; Arm C: Durvalumab + Rituximab ± Bendamustine
Drug: Ibrutinib — Administered orally
  Other Names: Imbruvica®
  Arms: Arm B: Durvalumab + Ibrutinib
Drug: Bendamustine — Administered as a 30-minute intravenous infusion
  Other Names: Treanda®; Bendeka®; Levact®
  Arms: Arm C: Durvalumab + Rituximab ± Bendamustine

SUMMARY:
This study is designed to determine the recommended phase 2 dose (RP2D), and the safety, and efficacy of durvalumab as monotherapy and when given in combination with lenalidomide and rituximab; ibrutinib; or bendamustine and rituximab at the RP2D in adults with lymphoma or chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
The study was to consist of 3 parts: dose-finding, dose-confirmation, and dose-expansion. In this study, 4 treatment arms were to be investigated:

* Arm A: durvalumab and lenalidomide ± rituximab
* Arm B: durvalumab and ibrutinib
* Arm C: durvalumab and rituximab ± bendamustine
* Arm D: durvalumab (monotherapy)

The study was to start with 3 dose-finding cohorts (Arms A, B, and C) and 1 dose-confirmation cohort (Arm D) in parallel. All treatment arms were to be open for enrollment at study start except in the US, where Arm D was to enroll depending on the availability of treatment slots and following the completion of assessment of responses from the combination therapy arms. For Arms A and C, prior to enrolling participants to receive all 3 drugs, the doublet combinations were to be evaluated. Once the doublet combinations were deemed tolerable, the eventual triplet combinations were to be tested.

On 05 September 2017, the US FDA issued a Partial Clinical Hold on the study Arm A. Following this Partial Clinical Hold no more participants were enrolled into study Arm A. Participants already enrolled and treated in Arm A who were receiving clinical benefit, based on the discretion of the investigator, could continue study treatment after being reconsented. Arm B and C completed dose confirmation. The dose expansion part of the study was not opened.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has histologically confirmed and documented B-cell lymphoma (eg, follicular, diffuse large B-cell, mantle cell, small lymphocytic, or Hodgkin lymphoma) and chronic lymphocytic leukemia.
2. Subject who has high-risk chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).
3. Subject who was previously treated with at least one prior systemic chemotherapy, immunotherapy, or chemoimmunotherapy.
4. Subject who has the Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
5. Subject who is willing and able to undergo biopsy.
6. Subject who has documented active relapsed or refractory disease requiring therapeutic intervention.
7. Subject with lymphoma who has measurable disease (≥ 2.0 cm in its longest dimension by computed tomography) or chronic lymphocytic leukemia in need of treatment.
8. Subject who fulfills the laboratory requirements as per protocol

Exclusion Criteria

1. Subject who has central nervous system (CNS) or meningeal involvement by lymphoma.
2. Subject who has any histopathologic finding consistent with myelodysplastic syndrome on bone marrow studies.
3. Subject who received any prior monoclonal antibodies against programmed cell death-1 (PD-1) or programmed cell death ligand-1 (PD-L1) and/or any prior:

   1. Arm A only: drugs with immunomodulatory and other properties (eg, lenalidomide, thalidomide);
   2. Arm B only: ibrutinib or other Bruton's tyrosine kinase (BTK) inhibitor;
   3. Arms C only: bendamustine
4. Subject who has active auto-immune disease.
5. Subject who has history of organ transplant or allogeneic hematopoietic stem cell transplantation.
6. Subject who is seropositive for or active viral infection with hepatitis B virus (HBV) (hepatitis B surface antigen [HBsAg] positive and/or detectable viral DNA)
7. Subject who has known seropositivity for or active infection for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
8. Subject who has history of primary immunodeficiency or tuberculosis.
9. Subject who other invasive malignancy within 2 years (5 years for Arm A) except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast, or incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) that has/have been surgically cured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2022-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (65):
- United States (18):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Shands Cancer Center University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Local Institution - 005, Rochester, New York
  - University of Rochester, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Jefferson Medical Oncology Associates, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
- France (13):
  - Centre Hospitalier Universitaire d'Avicennes, Bobigny
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier, Dijon
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - Local Institution - 102, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Local Institution - 105, Nantes
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Local Institution - 103, Pierre-Bénite
  - CHRU Rennes, Rennes
  - Centre Henri Becquerel, Rouen
- Germany (5):
  - Universitatsklinikum Essen, Essen
  - UKG Universitatsklinikum Gottingen, GÃ¶ttingen
  - Universitatsklinikum des Saarlandes, Homburg-Saar
  - Universitatsklinik Koln, KÃ¶ln
  - Medizinische Klinik III Klinikum der UniversitÃ¤t MÃ¼nchen-GroÃŸhadern, MÃ¼nchen
- Italy (9):
  - University of Bologna, Bologna
  - Local Institution - 306, Brescia
  - Spedali Civili Di Brescia, Brescia
  - IEO- Istituto Europeo di Oncologia, Milan
  - A.O. Ospedale Ca Granda - Niguarda, Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli, Campania
  - Local Institution - 304, Napoli, Campania
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - IRCCS Humanitas Clinical Institute, Rozzano (milano)
- Japan (4):
  - Local Institution - 602, Chuo-ku, Tokyo
  - National Cancer Center Hospital, Chūōku
  - Tokai University Hospital, Isehara City, Kanagawa
  - Aichi Cancer Center, Nagoya
- Netherlands (5):
  - VU Academic Medical Center, Amsterdam, Amsterdam
  - UMC Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medical Center, Rotterdam
  - Local Institution - 501, Rotterdam
- United Kingdom (11):
  - Local Institution - 402, Plymouth, Devon
  - Local Institution - 407, Nottingham, Nottinghamshire
  - St James University Hospital, Leeds
  - UCL Cancer Institute, London
  - Christie Hospital NHS Trust, Manchester
  - Local Institution - 404, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Local Institution - 406, Oxford
  - Oxford University Hospitals NHS Trust- Churchill Hospital-Oxford Centre for Respiratory Medicine, Oxford
  - Derriford Hospital, Plymouth
  - Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Derived] Casulo C, Santoro A, Cartron G, Ando K, Munoz J, Le Gouill S, Izutsu K, Rule S, Lugtenburg P, Ruan J, Arcaini L, Casadebaig ML, Fox B, Kilavuz N, Rettby N, Dell'Aringa J, Taningco L, Delarue R, Czuczman M, Witzig T. Durvalumab as monotherapy and in combination therapy in patients with lymphoma or chronic lymphocytic leukemia: The FUSION NHL 001 trial. Cancer Rep (Hoboken). 2023 Jan;6(1):e1662. doi: 10.1002/cnr2.1662. Epub 2022 Jul 19. PMID 35852004
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1, Arm A: DUR 1500 mg + LEN 20 mg: Participants received durvalumab (DUR) 1500 mg intravenous (IV) infusion on Day 1 of Cycles 1 through 13 (ie, 12 months) and lenalidomide (LEN) 20 mg orally once daily on Days 1 to 21 of Cycles 1 through 13 for participants with indolent non-Hodgkin's lymphoma (NHL) or for all cycles of treatment period until disease progression, unacceptable toxicity, or discontinuation for any other reason in participants with aggressive NHL.
- Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m²: Participants received durvalumab (DUR) 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and lenalidomide (LEN) 20 mg orally once daily on Days 1 to 21 of Cycles 1 through 13 for participants with indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in participants with aggressive NHL, and rituximab (RIT) 375 mg/m² IV infusion on Days 2, 8, 15, and 22 of Cycle 1 and on Day 1 of every 28-day cycle from Cycles 2 through 5.
- Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m²: Participants received durvalumab (DUR) 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and lenalidomide (LEN) 10 mg orally once daily on Days 1 to 21 of Cycles 1 through 13 for participants with indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in participants with aggressive NHL, and rituximab 375 mg/m² IV infusion on Days 2, 8, 15, 22 of Cycle 1 and on Day 1 of every 28-day cycle from Cycles 2 through 5.
- Part 1, Arm B: DUR 1500 mg + IBR 420 mg: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and ibrutinib (IBR) 420 mg orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
- Part 1, Arm B: DUR 1500 mg + IBR 560 mg: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and ibrutinib 560 mg orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
- Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m²: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6 (for participants with CLL the rituximab dose was 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose).
- Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m²: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and bendamustine (BEN) 70 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6.
- Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m²: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, bendamustine 70 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6 (for CLL the rituximab dose was 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose).
- Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m²: Participants received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, bendamustine 90 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6 (for CLL the rituximab dose was 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose).
- Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg: Participants with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and ibrutinib 420 mg orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
- Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg: Participants with mantle cell lymphoma (MCL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13 and ibrutinib 560 mg orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
- Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m²: Participants with follicular lymphoma (FL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, bendamustine 70 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6.
- Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m²: Participants with diffuse large B-cell lymphoma (DLBCL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, bendamustine 70 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6.
- Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m²: Participants with CLL or SLL received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13, bendamustine 70 mg/m² IV infusion on Days 1 and 2 of Cycles 1 through 6, and rituximab 375 mg/m² IV infusion on Day 2 of Cycles 1 through 6 (for CLL the rituximab dose was 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose).
- Part 2, Arm D FL: DUR 1500 mg: Participants with follicular lymphoma received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13.
- Part 2, Arm D DLBCL: DUR 1500 mg: Participants with diffuse large B-cell lymphoma (DLBCL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13.
- Part 2, Arm D CLL/SLL: DUR 1500 mg: Participants with CLL or SLL received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13.
- Part 2, Arm D MCL: DUR 1500 mg: Participants with mantle cell lymphoma (MCL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13.
- Part 2, Arm D HL: DUR 1500 mg: Participants with Hodgkin lymphoma (HL) received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 through 13.
Period: Overall Study
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Started | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 10 | 5 | 5 | 10 | 2 | 5 | 5
Participants Who Entered Follow-up Period After Completing/Discontinuing Study Treatment | 3 | 3 | 6 | 3 | 2 | 2 | 0 | 4 | 4 | 4 | 5 | 9 | 9 | 4 | 1 | 5 | 0 | 3 | 2
Completed | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 4 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not Completed | 3 | 2 | 7 | 3 | 3 | 3 | 1 | 3 | 5 | 4 | 6 | 6 | 9 | 4 | 5 | 10 | 2 | 5 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 2 | 1 | 3 | 1 | 2 | 3 | 0 | 3 | 3 | 2 | 2 | 2 | 8 | 1 | 4 | 7 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg | Total
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 10 | 5 | 5 | 10 | 2 | 5 | 5 | 106
Age, Continuous [Median (Full Range); unit: years] | 71.0 [50 to 78] | 66.0 [52 to 75] | 77.0 [53 to 80] | 58.0 [54 to 74] | 68.0 [57 to 81] | 79.0 [76 to 80] | 70.0 [70 to 70] | 68.0 [52 to 78] | 38.0 [21 to 77] | 68.0 [55 to 73] | 73.5 [54 to 84] | 64.5 [45 to 75] | 60.0 [46 to 71] | 68.0 [53 to 79] | 52.0 [39 to 71] | 61.5 [22 to 76] | 62.0 [55 to 69] | 77.0 [69 to 80] | 51.0 [34 to 65] | 67.0 [21 to 84]
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 3 | 4 | 2 | 5 | 7 | 2 | 3 | 5 | 1 | 0 | 4 | 44
  ≥ 65 Years | 2 | 2 | 6 | 1 | 3 | 3 | 1 | 3 | 2 | 6 | 8 | 5 | 3 | 3 | 2 | 5 | 1 | 5 | 1 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 3 | 3 | 1 | 3 | 4 | 2 | 2 | 4 | 1 | 2 | 2 | 35
  Male | 2 | 3 | 6 | 3 | 2 | 1 | 1 | 3 | 2 | 7 | 9 | 7 | 6 | 3 | 3 | 6 | 1 | 3 | 3 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 2 | 7 | 2 | 3 | 1 | 1 | 3 | 3 | 5 | 7 | 6 | 8 | 3 | 2 | 9 | 2 | 5 | 5 | 76
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 5 | 3 | 4 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 3 | 2 | 4 | 0 | 1 | 0 | 4 | 5 | 6 | 4 | 4 | 4 | 2 | 9 | 2 | 4 | 5 | 63
  Asian | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 13
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Collected or Reported | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 5 | 3 | 4 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 27
Histology [Count of Participants; unit: Participants]
  Follicular lymphoma | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 10 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 23
  Diffuse large B-cell lymphoma | 2 | 0 | 4 | 0 | 0 | 2 | 1 | 3 | 5 | 0 | 0 | 0 | 10 | 0 | 0 | 10 | 0 | 0 | 0 | 37
  Marginal zone lymphoma | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Transformed follicular lymphoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Mantle cell lymphoma | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 17
  CLL / SLL | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0 | 18
  Hodgkin lymphoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Eastern Cooperative Oncology Group ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: • 0 = Fully active, no restrictions; • 1 = Restricted activity but ambulatory, able to carry out work of a light nature; • 2 = Ambulatory and capable of all self-care but unable to carry out work activities; • 3 = Limited self-care, confined to bed or chair more than 50% of waking hours; • 4 = Completely disabled, no selfcare, confined to bed or chair; • 5 = Dead
  Participants
    0 - Fully Active | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 3 | 2 | 8 | 6 | 6 | 7 | 0 | 2 | 3 | 1 | 4 | 5 | 53
    1 - Restricted but ambulatory | 3 | 1 | 4 | 3 | 3 | 2 | 0 | 0 | 2 | 2 | 3 | 3 | 1 | 4 | 2 | 4 | 1 | 1 | 0 | 39
    2 - Ambulatory but unable to work | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 13
    3 - Limited self-care | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose limiting toxicities were evaluated during the DLT evaluation period for participants in the dose finding cohorts. The severity grading was determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03. A DLT is defined as below: Hematologic DLT • Grade 4 neutropenia observed for greater than 5 days duration • Grade 3 neutropenia associated with fever (≥ 38.5 °C) of any duration • Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding, or any requirement for platelets transfusion • Grade 4 anemia, unexplained by underlying disease • Any other grade 4 hematologic toxicity that does not resolve to participant's pretreatment baseline level within 72 hours. Non-Hematologic DLT • Any non-hematological toxicity ≥ Grade 3 except for alopecia and nausea controlled by medical management • Any treatment interruption greater than 2 weeks due to adverse event.
Time Frame: Cycle 1 (28 days)
Population: DLT Evaluable population included participants in Arms A, B, and C of Part 1, who took at least one dose of study drug and completed the DLT evaluation through the end of DLT evaluation period, or participants who took at least one dose of study drug and experienced at least one DLT prior to completion of the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m²
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 4 | 3 | 0 | 4 | 5
Participants | 0 | 3 | 1 | 0 | 0 | 0 |  | 0 | 1
Statistical Analysis 1: Comparison: Part 1, Arm B: DUR 1500 mg + IBR 420 mg vs Part 1, Arm B: DUR 1500 mg + IBR 560 mg; The safety review committee identified a preliminary recommended Phase 2 dose (RP2D) for each dose finding cohort based on an integrated assessment of the safety, pharmacokinetic, pharmacodynamic, and preliminary efficacy (as available); Test type: Other; For Arm B, ibrutinib 420 mg was confirmed as the RP2D for CLL/SLL participants and ibrutinib 560 mg was confirmed as the RP2D for MCL participants
Statistical Analysis 2: Comparison: Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² vs Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² vs Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² vs Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m²; [analysis description as in outcome 1, analysis 1]; Test type: Other; For Arm C the RP2D was confirmed as rituximab 375 mg/m² + bendamustine 70 mg/m²

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) occurring or worsening on or after the first dose of any study treatment (durvalumab, lenalidomide, ibrutinib, bendamustine or rituximab) and within 90 days after last dose of durvalumab or 28 days after the last dose of other study drugs, whichever was later, as well as those serious adverse events made known to the investigator at any time thereafter that were suspected of being related to study treatment. The intensity of AEs was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. For all other AEs not described in the CTCAE criteria, the intensity was assessed by the investigator as mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4), or death (Grade 5).
Time Frame: From first dose of any study drug to 90 days after last dose of durvalumab or 28 days after last dose of other study drugs, up to the data cut-off date of 6 March 2019. Maximum time on treatment was 55.4 weeks for DUR and 130 weeks for other study drugs.
Population: The Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 10 | 5 | 5 | 10 | 2 | 5 | 5
Participants
  Any TEAE | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 9 | 5 | 5 | 9 | 2 | 5 | 5
  TEAE Related to Any Study Drug | 3 | 3 | 8 | 3 | 4 | 3 | 0 | 4 | 5 | 10 | 9 | 10 | 9 | 5 | 4 | 3 | 0 | 3 | 2
  CTCAE Grade 3-4 TEAE | 1 | 3 | 7 | 2 | 3 | 2 | 1 | 3 | 4 | 8 | 10 | 6 | 9 | 5 | 4 | 7 | 1 | 4 | 3
  CTCAE Grade 3-4 TEAE Related to Any Study Drug | 1 | 3 | 7 | 1 | 1 | 2 | 0 | 2 | 2 | 7 | 6 | 5 | 7 | 3 | 3 | 2 | 0 | 1 | 1
  CTCAE Grade 5 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0
  CTCAE Grade 5 TEAE Related to Any Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAE | 1 | 2 | 4 | 2 | 2 | 2 | 1 | 1 | 3 | 6 | 7 | 5 | 5 | 2 | 4 | 7 | 0 | 3 | 2
  Serious TEAE Related to Any Study Drug | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 3 | 3 | 1 | 3 | 1 | 0 | 0 | 0
  TEAE Leading to Discontinuation of Any Study Drug | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0
  TEAE Leading to Dose Modifications of Study Drug | 1 | 3 | 3 | 3 | 4 | 3 | 1 | 4 | 4 | 8 | 9 | 7 | 4 | 3 | 2 | 0 | 0 | 3 | 3

3. Secondary Outcome: Overall Response Rate (ORR) During Durvalumab Treatment
Description: For lymphoma participants, response evaluation was based on International Working Group (IWG) response criteria for malignant lymphoma (the Lugano Classification). Overall response rate is defined as the percent of participants with best response of complete response (CR) or partial response (PR). For chronic lymphocytic leukemia participants, response evaluation was based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines for diagnosis and treatment of CLL. The ORR is defined as the percent of participants with best response of CR, complete response with incomplete marrow recovery (CRi), nodular partial response (nPR), PR, or partial response with lymphocytosis (PRL).
Time Frame: Up to 13 cycles (12 months)
Population: The Efficacy Evaluable population includes all participants who completed at least 1 cycle of their assigned treatment, and have baseline and at least 1 post-baseline tumor response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 4 | 3 | 0 | 4 | 4 | 9 | 10 | 9 | 10 | 4 | 5 | 10 | 2 | 5 | 5
percentage of participants | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 75.0 [19.4 to 99.4] | 33.3 [0.8 to 90.6] |  | 50.0 [6.8 to 93.2] | 0 [NA to NA] — Not calculated for zero responses | 88.9 [51.8 to 99.7] | 60.0 [26.2 to 87.8] | 88.9 [51.8 to 99.7] | 30.0 [6.7 to 65.2] | 50.0 [6.8 to 93.2] | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 20.0 [0.5 to 71.6]

4. Secondary Outcome: Overall Response Rate During the Entire Study
Description: For lymphoma participants, response evaluation was based on International Working Group (IWG) response criteria for malignant lymphoma (the Lugano Classification) (Cheson, 2014). Overall response rate is defined as the percent of participants with best response of complete response (CR) or partial response (PR). For chronic lymphocytic leukemia participants, response evaluation was based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines for diagnosis and treatment of CLL. The ORR is defined as the percentage of participants with best response of CR, complete response with incomplete marrow recovery (CRi), nodular partial response (nPR), PR, or partial response with lymphocytosis (PRL).
Time Frame: From first dose of any study drug to the end of follow-up, up to the data cutoff date of March 6, 2019; median (minimum, maximum) time on study was 16.7 (0.9, 32.9) months.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 4 | 3 | 0 | 4 | 4 | 9 | 10 | 9 | 10 | 4 | 5 | 10 | 2 | 5 | 5
percentage of participants | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 75.0 [19.4 to 99.4] | 33.3 [0.8 to 90.6] |  | 50.0 [6.8 to 93.2] | 0 [NA to NA] — Not calculated for zero responses | 100.0 [66.4 to 100.0] | 70.0 [34.8 to 93.3] | 88.9 [51.8 to 99.7] | 30.0 [6.7 to 65.2] | 50.0 [6.8 to 93.2] | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 0 [NA to NA] — Not calculated for zero responses | 20.0 [0.5 to 71.6]

5. Secondary Outcome: Time to First Response
Description: Time to response was calculated as the time from first dose of study drug to the first response date (CR or PR for lymphoma participants and CR, CRi, nPR, PR, or PRL for CLL participants).
Time Frame: as for outcome 4
Population: Efficacy evaluable population (all participants who completed at least 1 cycle of their assigned treatment, and have baseline and at least 1 post-baseline tumor response assessment) who had an objective response
Measure: Median (Full Range); unit: weeks
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 2 | 2 | 4 | 2 | 3 | 1 | 0 | 2 | 0 | 9 | 7 | 8 | 3 | 2 | 0 | 0 | 0 | 0 | 1
weeks | 70.85 [12.1 to 129.6] | 12.60 [12.1 to 13.1] | 18.20 [11.3 to 36.1] | 11.85 [11.4 to 12.3] | 13.40 [12.4 to 52.9] | 13.00 [13.0 to 13.0] |  | 13.10 [12.1 to 14.1] |  | 12.10 [10.9 to 72.9] | 12.10 [6.6 to 26.4] | 12.35 [10.3 to 15.3] | 12.00 [8.7 to 12.1] | 12.10 [12.1 to 12.1] |  |  |  |  | 13.10 [13.1 to 13.1]

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response
Description: Duration of response is defined for responders only as the time from the first documented response (CR or PR for lymphoma participants or CR, CRi, nPR, PR, or PRL for CLL participants) to disease progression or death (from any cause). For participants with response but no progression, or death, duration of response was censored at the last date that the participant was known to be progression-free.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 2 | 2 | 4 | 2 | 3 | 1 | 0 | 2 | 0 | 9 | 7 | 8 | 3 | 2 | 0 | 0 | 0 | 0 | 1
weeks | 10.14 [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | 29.29 [NA to NA] — Could not be evaluated due to the low number of events |  | NA [NA to NA] — Could not be evaluated due to the low number of events |  | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | 24.14 [9.14 to 26.14] | NA [NA to NA] — Could not be evaluated due to the low number of events |  |  |  |  | 11.14 [NA to NA] — Could not be evaluated due to the low number of events

7. Secondary Outcome: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: Progression-free survival was calculated as the time from first dose of study drug to the first documented progression or death (from any cause) during the entire efficacy evaluation period. For participants with no progression or death, PFS was censored at the last assessment date the participant was known to be progression-free.
Time Frame: as for outcome 4
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 10 | 5 | 5 | 10 | 2 | 5 | 5
months | 8.41 [5.09 to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | 28.71 [4.50 to NA] — Could not be evaluated due to the low number of events | 9.69 [1.64 to 12.68] | 1.25 [NA to NA] — Could not be evaluated due to the low number of events | 3.82 [1.25 to NA] — Could not be evaluated due to the low number of events | 2.48 [0.49 to 5.91] | NA [NA to NA] — Could not be evaluated due to the low number of events | NA [NA to NA] — Could not be evaluated due to the low number of events | 14.65 [5.75 to 14.65] | 2.06 [0.76 to 8.28] | NA [NA to NA] — Could not be evaluated due to the low number of events | 1.68 [0.69 to 4.63] | 1.17 [0.26 to 3.19] | 2.76 [2.50 to 3.02] | 2.33 [0.79 to 10.02] | 2.66 [2.56 to 5.98]

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Durvalumab
Time Frame: Cycle 1, Day 1 (pre-dose and at end of infusion), and 4, 24, 48, 168 (Day 8), 336 (Day 15), and 508 (Day 22) hours after the end of infusion.
Population: The Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Groups:
- Arm A: Durvalumab + Lenalidomide ± Rituximab: Participants assigned to Arm A received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, and 10 mg or 20 mg lenalidomide orally once daily on Days 1 to 21 of Cycles 1 to 13 in indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in aggressive NHL, and rituximab 375 mg/m² IV weekly in Cycle 1 and on Day 1 of Cycles 2 to 5.
- Arm B: Durvalumab + Ibrutinib: Participants assigned to Arm B received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, and 420 or 560 mg ibrutinib orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason.
- Arm C: Durvalumab + Bendamustine ± Rituximab: Participants assigned to Arm C received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, 70 or 90 mg/m² bendamustine IV on Days 1 and 2 of Cycles 1 to 6, and rituximab 375 mg/m² IV on Day 2 of Cycles 1 to 6 (for CLL the rituximab dose was 375 mg/m² Cycle 1 first dose and 500 mg/m² for each subsequent dose).
- Arm D: Durvalumab Monotherapy: Participants assigned to Arm D received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13.
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 26
μg/L | 420264.066 (22.7) | 361906.229 (30.1) | 331572.478 (33.4) | 392663.668 (41.1)

9. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Durvalumab
Time Frame: as for outcome 8
Population: PK population
Measure: Median (Full Range); unit: days
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 26
days | 0.0510 [0.042 to 1.035] | 0.0479 [0.041 to 1.061] | 0.0510 [0.042 to 6.788] | 0.0420 [0.038 to 1.986]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUClast) of Durvalumab
Time Frame: as for outcome 8
Population: The PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*μg/L
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 26
days*μg/L | 3120149.759 (29.5) | 3225869.344 (31.9) | 2670168.397 (46.7) | 3053060.746 (37.8)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Durvalumab
Time Frame: as for outcome 8
Population: The PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*μg/L
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 25
days*μg/L | 4867431.378 (23.3) | 5818262.846 (42.1) | 4762968.345 (71.0) | 5593532.553 (53.0)

12. Secondary Outcome: Terminal Elimination Phase Half-Life (t½) of Durvalumab
Time Frame: as for outcome 8
Population: The PK population
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: days
Groups:
- Arm A: Durvalumab + Lenalidomide Â± Rituximab: Participants assigned to Arm A received durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, and 10 mg or 20 mg lenalidomide orally once daily on Days 1 to 21 of Cycles 1 to 13 in indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in aggressive NHL, and rituximab 375 mg/m² IV weekly in Cycle 1 and on Day 1 of Cycles 2 to 5.
Arm/Group | Arm A: Durvalumab + Lenalidomide Â± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 25
days | 11.596 (46.6) | 17.344 (47.3) | 16.327 (57.4) | 15.399 (53.5)

13. Secondary Outcome: Clearance (CL) of Durvalumab
Time Frame: as for outcome 8
Population: The PK population
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 25
L/day | 0.3082 (23.3) | 0.2578 (42.1) | 0.3149 (71.0) | 0.2682 (53.0)

14. Secondary Outcome: Volume of Distribution (Vz) of Durvalumab
Time Frame: as for outcome 8
Population: The PK population
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Arm A: Durvalumab + Lenalidomide ± Rituximab | Arm B: Durvalumab + Ibrutinib | Arm C: Durvalumab + Bendamustine ± Rituximab | Arm D: Durvalumab Monotherapy
Number analyzed (Participants) | 14 | 27 | 38 | 25
liters | 5.155 (41.9) | 6.451 (38.3) | 7.418 (33.7) | 5.957 (33.0)

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lenalidomide
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, and 24 hours post-dose, and Cycle 1 Day 15 at pre-dose, 1, 2, and 4 hours post-dose.
Population: PK population with available data at each time point
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Arm A: Lenalidomide 10 mg: Participants in Arm A received lenalidomide 10 mg orally once daily on Days 1 to 21 of Cycles 1 to 13 for participants with indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in participants with aggressive NHL, and durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, and rituximab 375 mg/m² IV weekly in Cycle 1 and on Day 1 of Cycles 2 to 5.
- Arm A: Lenalidomide 20 mg: Participants in Arm A received lenalidomide 20 mg orally once daily on Days 1 to 21 of Cycles 1 to 13 for participants with indolent NHL or until disease progression, unacceptable toxicity, or discontinuation for any other reason in participants with aggressive NHL, and durvalumab 1500 mg IV infusion on Day 1 of Cycles 1 to 13, and rituximab 375 mg/m² IV weekly in Cycle 1 and on Day 1 of Cycles 2 to 5.
Arm/Group | Arm A: Lenalidomide 10 mg | Arm A: Lenalidomide 20 mg
Number analyzed (Participants) | 5 | 4
ng/mL
  Cycle 1 Day 1 | 141.881 (22.0) | 309.917 (6.9)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 1
  Cycle 1 Day 15 | 107.635 (40.9) | 174.090

16. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Lenalidomide
Time Frame: as for outcome 15
Population: PK population with available data at each time point
Measure: Median (Full Range); unit: hours
Arm/Group | Arm A: Lenalidomide 10 mg | Arm A: Lenalidomide 20 mg
Number analyzed (Participants) | 5 | 4
hours
  Cycle 1 Day 1 | 1.9500 [1.000 to 3.917] | 1.1667 [1.000 to 1.433]
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 1
  Cycle 1 Day 15 | 3.0333 [1.233 to 4.000] | 1.000 [1.000 to 1.000]

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUClast) of Lenalidomide
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, and 24 hours post-dose
Population: PK population with available data
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Arm A: Lenalidomide 10 mg | Arm A: Lenalidomide 20 mg
Number analyzed (Participants) | 5 | 4
h*ng/mL | 789.297 (84.3) | 805.299 (56.0)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ibrutinib
Time Frame: as for outcome 15
Population: PK population with available data at each time point
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Arm B: Ibrutinib 420 mg: Participants assigned to Arm B received 420 mg ibrutinib orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason, and durvalumab 1500 mg IV on Day 1 of Cycles 1 to 13.
- Arm B: Ibrutinib 560 mg: Participants assigned to Arm B received 560 mg ibrutinib orally once daily until disease progression, unacceptable toxicity or discontinuation for any other reason, and durvalumab 1500 mg IV on Day 1 of Cycles 1 to 13.
Arm/Group | Arm B: Ibrutinib 420 mg | Arm B: Ibrutinib 560 mg
Number analyzed (Participants) | 13 | 13
ng/mL
  Cycle 1 Day 1 | 129.704 (98.0) | 67.728 (197.9)
  Cycle 1 Day 15: number analyzed (Participants) | 9 | 10
  Cycle 1 Day 15 | 86.840 (136.9) | 72.436 (166.3)

19. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Ibrutinib
Time Frame: as for outcome 15
Population: PK population with available data at each time point
Measure: Median (Full Range); unit: hours
Arm/Group | Arm B: Ibrutinib 420 mg | Arm B: Ibrutinib 560 mg
Number analyzed (Participants) | 13 | 13
hours
  Cycle 1 Day 1 | 2.000 [0.000 to 4.367] | 1.9333 [0.933 to 3.917]
  Cycle 1 Day 15: number analyzed (Participants) | 9 | 10
  Cycle 1 Day 15 | 1.8833 [1.000 to 4.000] | 2.000 [1.000 to 4.083]

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUClast) of Ibrutinib
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, and 24 hours post-dose
Population: PK population with available data
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Arm B: Ibrutinib 420 mg | Arm B: Ibrutinib 560 mg
Number analyzed (Participants) | 13 | 13
h*ng/mL | 586.396 (117.2) | 436.855 (246.5)

21. Secondary Outcome: Change From Baseline in Soluble Programmed Cell Death Ligand-1 (sPD-L1) Concentration
Description: Change from baseline in sPD-L1 could not be calculated as all post-baseline samples were below the lower limit of quantification (<15.60 pg/mL).
Time Frame: Baseline (Cycle 1 Day 1 predose) and Day 1 of Cycles 2 to 13
Population: Biomarker Evaluable Population included all participants who received at least 1 dose of study drug and had at least 1 non-missing biomarker assessment. No participants had quantifiable sPD-L1 measurements post-baseline.
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Post Hoc Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) - Extended Collection
Description: TEAEs defined as AEs occurring or worsening on or after first dose of any study treatment (durvalumab, lenalidomide, ibrutinib, bendamustine or rituximab) and within 90 days after last dose of durvalumab or 28 days after the last dose of other study drugs, whichever was later, as well as those serious adverse events made known to the investigator at any time thereafter that were suspected of being related to study treatment. Intensity of AEs graded according to the NCI CTCAE V. 4.03. For all other AEs not described in the CTCAE criteria, the intensity was assessed by investigator as mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4), or death (Grade 5). This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date (assessments made until August 21, 2022).
Time Frame: From first dose of any study drug to 90 days after last dose of durvalumab or 28 days after last dose of other study drugs, up to the study completion date of August 21, 2022 (up to approximately 75 months).
Population: The Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 10 | 5 | 5 | 10 | 2 | 5 | 5
Participants
  Any TEAE | 3 | 3 | 8 | 3 | 4 | 3 | 1 | 4 | 5 | 10 | 10 | 10 | 9 | 5 | 5 | 9 | 2 | 5 | 5
  TEAE Related to Any Study Drug | 3 | 3 | 8 | 3 | 4 | 3 | 0 | 4 | 5 | 10 | 9 | 10 | 9 | 5 | 4 | 3 | 0 | 3 | 2
  CTCAE Grade 3-4 TEAE | 1 | 3 | 7 | 2 | 4 | 2 | 1 | 3 | 4 | 9 | 10 | 6 | 9 | 5 | 4 | 7 | 1 | 4 | 3
  CTCAE Grade 3-4 TEAE Related to Any Study Drug | 1 | 3 | 7 | 1 | 1 | 2 | 0 | 2 | 2 | 8 | 6 | 5 | 7 | 3 | 3 | 2 | 0 | 1 | 1
  CTCAE Grade 5 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0
  CTCAE Grade 5 TEAE Related to Any Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAE | 1 | 2 | 4 | 2 | 3 | 2 | 1 | 1 | 3 | 6 | 7 | 5 | 5 | 2 | 4 | 7 | 0 | 3 | 2
  Serious TEAE Related to Any Study Drug | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 3 | 3 | 1 | 3 | 1 | 0 | 0 | 0
  TEAE Leading to Discontinuation of Any Study Drug | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0
  TEAE Leading to Dose Modifications of Study Drug | 1 | 3 | 5 | 3 | 4 | 3 | 1 | 4 | 4 | 9 | 9 | 7 | 4 | 3 | 2 | 0 | 0 | 3 | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from the participants first dose to their study completion (up to approximately 75 months). SAEs and Other AEs were assessed from first dose to 90 days from the last dose of durvalumab or 28 days from the last dose of any other study treatment [ie, lenalidomide, ibrutinib, rituximab, bendamustine, or involved field radiation (IFRT) therapy], whichever occurs later (up to approximately 75 months).
Arm/Group | Part 1, Arm A: DUR 1500 mg + LEN 20 mg | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² | Part 1, Arm B: DUR 1500 mg + IBR 420 mg | Part 1, Arm B: DUR 1500 mg + IBR 560 mg | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² | Part 2, Arm D FL: DUR 1500 mg | Part 2, Arm D DLBCL: DUR 1500 mg | Part 2, Arm D CLL/SLL: DUR 1500 mg | Part 2, Arm D MCL: DUR 1500 mg | Part 2, Arm D HL: DUR 1500 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 2/8 | 0/3 | 3/4 | 2/3 | 1/1 | 3/4 | 4/5 | 1/10 | 2/10 | 0/10 | 9/10 | 2/5 | 4/5 | 9/10 | 0/2 | 4/5 | 4/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 4/8 | 2/3 | 3/4 | 2/3 | 1/1 | 1/4 | 3/5 | 6/10 | 7/10 | 5/10 | 5/10 | 2/5 | 4/5 | 8/10 | 0/2 | 4/5 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 3/3 | 4/4 | 3/3 | 1/1 | 4/4 | 5/5 | 10/10 | 10/10 | 10/10 | 9/10 | 5/5 | 5/5 | 10/10 | 2/2 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Arm A: DUR 1500 mg + LEN 20 mg (N=3) | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² (N=3) | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² (N=8) | Part 1, Arm B: DUR 1500 mg + IBR 420 mg (N=3) | Part 1, Arm B: DUR 1500 mg + IBR 560 mg (N=4) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² (N=3) | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² (N=1) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=4) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² (N=5) | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg (N=10) | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg (N=10) | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=10) | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=10) | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=5) | Part 2, Arm D FL: DUR 1500 mg (N=5) | Part 2, Arm D DLBCL: DUR 1500 mg (N=10) | Part 2, Arm D CLL/SLL: DUR 1500 mg (N=2) | Part 2, Arm D MCL: DUR 1500 mg (N=5) | Part 2, Arm D HL: DUR 1500 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Arm A: DUR 1500 mg + LEN 20 mg (N=3) | Part 1, Arm A: DUR 1500 mg + LEN 20 mg + RIT 375 mg/m² (N=3) | Part 1, Arm A: DUR 1500 mg + LEN 10 mg + RIT 375 mg/m² (N=8) | Part 1, Arm B: DUR 1500 mg + IBR 420 mg (N=3) | Part 1, Arm B: DUR 1500 mg + IBR 560 mg (N=4) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² (N=3) | Part 1, Arm C: DUR 1500 mg + BEN 70 mg/m² (N=1) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=4) | Part 1, Arm C: DUR 1500 mg + RIT 375 mg/m² + BEN 90 mg/m² (N=5) | Part 2, Arm B CLL/SLL: DUR 1500 mg + IBR 420 mg (N=10) | Part 2, Arm B MCL: DUR 1500 mg + IBR 560 mg (N=10) | Part 2, Arm C FL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=10) | Part 2 Arm C DLBCL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=10) | Part 2, Arm C CLL/SLL: DUR 1500 mg + RIT 375 mg/m² + BEN 70 mg/m² (N=5) | Part 2, Arm D FL: DUR 1500 mg (N=5) | Part 2, Arm D DLBCL: DUR 1500 mg (N=10) | Part 2, Arm D CLL/SLL: DUR 1500 mg (N=2) | Part 2, Arm D MCL: DUR 1500 mg (N=5) | Part 2, Arm D HL: DUR 1500 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 3 | 1 | 5 | 1 | 1 | 2 | 2 | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1 | 1 | 1 | 0 | 2 | 1 | 4 | 3 | 6 | 3 | 1 | 0 | 3 | 2 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 3 | 3 | 2 | 6 | 1 | 1 | 4 | 2 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epidermolysis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 1 | 5 | 5 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 3 | 2 | 1 | 1 | 0 | 3 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 2 | 3 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 3 | 3 | 2 | 3 | 4 | 1 | 2 | 6 | 1 | 4 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunodeficiency (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 2 | 2 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 1 | 4 | 2 | 1 | 2 | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 2 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 4 | 4 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gravitational oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumatosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stenotrophomonas sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint noise (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was placed on full clinical hold by the United States (US) Food and Drug Administration (FDA) on 05 Sep 2017. As the result, the study was closed for further enrollment, and all participants were discontinued from all study treatments (durvalumab, lenalidomide and dexamethasone). All participants were followed for second primary malignancies (SPMs) for 5 years after the last participant has been enrolled as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (3):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02733042/Prot_003.pdf
  • Statistical Analysis Plan: MEDI4736-NHL-001_SAP_Redacted.14Dec2017 (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02733042/SAP_001.pdf
  • Statistical Analysis Plan: MEDI4736-NHL-001_SAP_Amendment_1_Redacted.14Dec2017 (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02733042/SAP_002.pdf